CLINICAL TRIAL: NCT04024410
Title: Optimal Positive End-expiratory Pressure (PEEP) in Prone Position During Spine Surgery. A Prospective Observational Study
Brief Title: Optimal Positive End-expiratory Pressure (PEEP) in Prone Position During Spine Surgery
Acronym: OPTIPRONE
Status: Completed | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/8270/I
Record Dates: First submitted 2019-06-27; First posted 2019-07-18 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2019-06

CONDITIONS: Anesthesia; Surgery
Keywords: prone position; anesthesia, general; end-expiratory pressure, positive; respiration, artificial
MeSH Terms: conditions — Respiratory Aspiration | interventions — Prone Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluation of PEEP in prone position — Assessment of optimal Positive End-Expiratory Pressure (PEEP) in patients undergoing scheduled spine surgery in prone position.

SUMMARY:
Background:

There is a lack of studies regarding Optimal (best) positive end-expiratory pressure (PEEP) in prone position during surgery, and its relation with optimal PEEP in supine position.

Hypothesis:

In patients undergoing scheduled spinal surgery, optimal PEEP in the prone position is lower than optimal PEEP in the supine position.

Aims:

To assess the difference optimal PEEP in supine vs. prone positions in patients undergoing spine surgery.

To evaluate the changes in optimal PEEP in prone position throughout the surgical procedure.

Methods:

Observational study, one center. Main variable: optimal PEEP. Secondary variables: PaO2, pCO2 and dynamic compliance (Crd) in prone and supine position.

DETAILED DESCRIPTION:
Recruitment: Patients scheduled for spine surgery were Main outcome: Optimal PEEP determined after a pulmonary recruitment manoeuvre in supine and in prone position and every hour during the surgery in prone position.

Secondary outcomes: Pulmonary compliance, blood gas analysis and hemodynamic parameters

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Spine prone surgery lasting ≥2 hours.
* Absence of known pulmonary pathology.

Exclusion Criteria:

* Pregnancy or lactation.
* Contraindication to alveolar recruitment maneuvers (risk of barotrauma, hemodynamic instability).
* Body mass index (BMI) >35.
* Heart failure defined as IC <2.5 L/min/m2 and/or inotropic support requirements prior to surgery.
* Diagnosis or suspicion of intracranial hypertension (intracranial pressure >15 mmHg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for spine surgery that requires prone decubitus.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

PRIMARY OUTCOMES:
Positive End-Expiratory Pressure (PEEP) | 10 minutes after intubation
  Positive End-Expiratory Pressure (cmH2O) in supine position
Positive End-Expiratory Pressure (PEEP) | 10 minutes after positioning
  Positive End-Expiratory Pressure (cmH2O) in prone position
Change in Positive End-Expiratory Pressure (PEEP) | From determination of optimal PEEP until the first hour and then every hour, assessed up to the end of surgery (maximum 6 hours)
  Variation of Positive End-Expiratory Pressure (cmH2O) during surgery in prone position with respect to PEEP value at 10 minutes after positioning

SECONDARY OUTCOMES:
Static compliance | 10 minutes after intubation
  Tidal volume / Plateau pressure ratio (mL/cmH2O) in supine position
Static compliance | 10 minutes after positioning
  Tidal volume / Plateau pressure ratio (mL/cmH2O) in prone position
Change in static compliance | Measured at the same time as Auto PEEP until the first hour and then every hour, assessed up to the end of surgery (maximum 6 hours)
  Variation of static compliance (Tidal volume / Plateau pressure ratio, in mL/cmH2O) during surgery in prone position
Arterial oxygen pressure (PaO2) | 10 minutes after intubation
  Partial pressure of oxygen (mmHg) in supine position
Arterial oxygen pressure (PaO2) | 10 minutes after positioning
  Partial pressure of oxygen (mmHg) in prone position
Change in arterial oxygen pressure (PaO2) | Measured at the same time as Auto PEEP until the first hour and then every hour, assessed up to the end of surgery (maximum 6 hours)
  Variation of partial pressure of oxygen (mmHg) during surgery in prone position
Arterial carbon dioxide pressure (PaCO2) | 10 minutes after intubation
  Partial pressure of carbon dioxide (mmHg) in supine position
Arterial carbon dioxide pressure (PaCO2) | 10 minutes after positioning
  Partial pressure of carbon dioxide (mmHg) in prone position
Change in arterial carbon dioxide pressure (PaCO2) | Measured at the same time as Auto PEEP until the first hour and then every hour, assessed up to the end of surgery (maximum 6 hours)
  Variation of partial pressure of carbon dioxide (mmHg) during surgery in prone position

CONTACTS AND LOCATIONS:
Overall Officials: Lluís Gallart, Dr, Principal Investigator — Hospital del Mar (Barcelona, Spain)
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Slutsky AS, Ranieri VM. Ventilator-induced lung injury. N Engl J Med. 2013 Nov 28;369(22):2126-36. doi: 10.1056/NEJMra1208707. No abstract available. PMID 24283226
- [Background] Canet J, Gallart L, Gomar C, Paluzie G, Valles J, Castillo J, Sabate S, Mazo V, Briones Z, Sanchis J; ARISCAT Group. Prediction of postoperative pulmonary complications in a population-based surgical cohort. Anesthesiology. 2010 Dec;113(6):1338-50. doi: 10.1097/ALN.0b013e3181fc6e0a. PMID 21045639
- [Background] Serpa Neto A, Cardoso SO, Manetta JA, Pereira VG, Esposito DC, Pasqualucci Mde O, Damasceno MC, Schultz MJ. Association between use of lung-protective ventilation with lower tidal volumes and clinical outcomes among patients without acute respiratory distress syndrome: a meta-analysis. JAMA. 2012 Oct 24;308(16):1651-9. doi: 10.1001/jama.2012.13730. PMID 23093163
- [Background] Duggan M, Kavanagh BP. Pulmonary atelectasis: a pathogenic perioperative entity. Anesthesiology. 2005 Apr;102(4):838-54. doi: 10.1097/00000542-200504000-00021. PMID 15791115
- [Background] Goldenberg NM, Steinberg BE, Lee WL, Wijeysundera DN, Kavanagh BP. Lung-protective ventilation in the operating room: time to implement? Anesthesiology. 2014 Jul;121(1):184-8. doi: 10.1097/ALN.0000000000000274. No abstract available. PMID 24781494
- [Background] Futier E, Constantin JM, Paugam-Burtz C, Pascal J, Eurin M, Neuschwander A, Marret E, Beaussier M, Gutton C, Lefrant JY, Allaouchiche B, Verzilli D, Leone M, De Jong A, Bazin JE, Pereira B, Jaber S; IMPROVE Study Group. A trial of intraoperative low-tidal-volume ventilation in abdominal surgery. N Engl J Med. 2013 Aug 1;369(5):428-37. doi: 10.1056/NEJMoa1301082. PMID 23902482
- [Background] Coppola S, Froio S, Chiumello D. Protective lung ventilation during general anesthesia: is there any evidence? Crit Care. 2014 Mar 18;18(2):210. doi: 10.1186/cc13777. No abstract available. PMID 25029254
- [Background] Ladha K, Vidal Melo MF, McLean DJ, Wanderer JP, Grabitz SD, Kurth T, Eikermann M. Intraoperative protective mechanical ventilation and risk of postoperative respiratory complications: hospital based registry study. BMJ. 2015 Jul 14;351:h3646. doi: 10.1136/bmj.h3646. PMID 26174419
- [Background] Hemmes SN, Serpa Neto A, Schultz MJ. Intraoperative ventilatory strategies to prevent postoperative pulmonary complications: a meta-analysis. Curr Opin Anaesthesiol. 2013 Apr;26(2):126-33. doi: 10.1097/ACO.0b013e32835e1242. PMID 23385321
- [Background] Hemmes SN, Severgnini P, Jaber S, Canet J, Wrigge H, Hiesmayr M, Tschernko EM, Hollmann MW, Binnekade JM, Hedenstierna G, Putensen C, de Abreu MG, Pelosi P, Schultz MJ. Rationale and study design of PROVHILO - a worldwide multicenter randomized controlled trial on protective ventilation during general anesthesia for open abdominal surgery. Trials. 2011 May 6;12:111. doi: 10.1186/1745-6215-12-111. PMID 21548927
- [Background] Gattinoni L, Caironi P. Prone positioning: beyond physiology. Anesthesiology. 2010 Dec;113(6):1262-4. doi: 10.1097/ALN.0b013e3181fcd97e. No abstract available. PMID 21042196
- [Background] Pelosi P, Caironi P, Taccone P, Brazzi L. Pathophysiology of prone positioning in the healthy lung and in ALI/ARDS. Minerva Anestesiol. 2001 Apr;67(4):238-47. PMID 11376516
- [Background] Edgcombe H, Carter K, Yarrow S. Anaesthesia in the prone position. Br J Anaesth. 2008 Feb;100(2):165-83. doi: 10.1093/bja/aem380. PMID 18211991
- [Background] Mure M, Domino KB, Lindahl SG, Hlastala MP, Altemeier WA, Glenny RW. Regional ventilation-perfusion distribution is more uniform in the prone position. J Appl Physiol (1985). 2000 Mar;88(3):1076-83. doi: 10.1152/jappl.2000.88.3.1076. PMID 10710406
- [Background] Pelosi P, Croci M, Calappi E, Cerisara M, Mulazzi D, Vicardi P, Gattinoni L. The prone positioning during general anesthesia minimally affects respiratory mechanics while improving functional residual capacity and increasing oxygen tension. Anesth Analg. 1995 May;80(5):955-60. doi: 10.1097/00000539-199505000-00017. PMID 7726438
- [Background] Pelosi P, Croci M, Calappi E, Mulazzi D, Cerisara M, Vercesi P, Vicardi P, Gattinoni L. Prone positioning improves pulmonary function in obese patients during general anesthesia. Anesth Analg. 1996 Sep;83(3):578-83. doi: 10.1097/00000539-199609000-00025. PMID 8780285
- [Background] Petersson J, Ax M, Frey J, Sanchez-Crespo A, Lindahl SG, Mure M. Positive end-expiratory pressure redistributes regional blood flow and ventilation differently in supine and prone humans. Anesthesiology. 2010 Dec;113(6):1361-9. doi: 10.1097/ALN.0b013e3181fcec4f. PMID 21068656
- [Background] Beitler JR, Guerin C, Ayzac L, Mancebo J, Bates DM, Malhotra A, Talmor D. PEEP titration during prone positioning for acute respiratory distress syndrome. Crit Care. 2015 Dec 21;19:436. doi: 10.1186/s13054-015-1153-9. PMID 26686509
- [Background] Fan E, Del Sorbo L, Goligher EC, Hodgson CL, Munshi L, Walkey AJ, Adhikari NKJ, Amato MBP, Branson R, Brower RG, Ferguson ND, Gajic O, Gattinoni L, Hess D, Mancebo J, Meade MO, McAuley DF, Pesenti A, Ranieri VM, Rubenfeld GD, Rubin E, Seckel M, Slutsky AS, Talmor D, Thompson BT, Wunsch H, Uleryk E, Brozek J, Brochard LJ; American Thoracic Society, European Society of Intensive Care Medicine, and Society of Critical Care Medicine. An Official American Thoracic Society/European Society of Intensive Care Medicine/Society of Critical Care Medicine Clinical Practice Guideline: Mechanical Ventilation in Adult Patients with Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2017 May 1;195(9):1253-1263. doi: 10.1164/rccm.201703-0548ST. PMID 28459336
- [Background] Spaeth J, Daume K, Goebel U, Wirth S, Schumann S. Increasing positive end-expiratory pressure (re-)improves intraoperative respiratory mechanics and lung ventilation after prone positioning. Br J Anaesth. 2016 Jun;116(6):838-46. doi: 10.1093/bja/aew115. PMID 27199315
- [Background] Katoh T, Suguro Y, Ikeda T, Kazama T, Ikeda K. Influence of age on awakening concentrations of sevoflurane and isoflurane. Anesth Analg. 1993 Feb;76(2):348-52. PMID 8424514
- [Background] Pelosi P, Gama de Abreu M, Rocco PR. New and conventional strategies for lung recruitment in acute respiratory distress syndrome. Crit Care. 2010;14(2):210. doi: 10.1186/cc8851. Epub 2010 Mar 9. PMID 20236454
- [Background] Ferrando C, Mugarra A, Gutierrez A, Carbonell JA, Garcia M, Soro M, Tusman G, Belda FJ. Setting individualized positive end-expiratory pressure level with a positive end-expiratory pressure decrement trial after a recruitment maneuver improves oxygenation and lung mechanics during one-lung ventilation. Anesth Analg. 2014 Mar;118(3):657-65. doi: 10.1213/ANE.0000000000000105. PMID 24557111
- [Background] Mahajan RP, Hennessy N, Aitkenhead AR, Jellinek D. Effect of three different surgical prone positions on lung volumes in healthy volunteers. Anaesthesia. 1994 Jul;49(7):583-6. doi: 10.1111/j.1365-2044.1994.tb14224.x. PMID 8042721